CLINICAL TRIAL: NCT00621049
Title: Randomized Phase II Trial of Adjuvant Carboplatin, Docetaxel, Bevacizumab, and Erlotinib Versus Chemotherapy Alone in Patients With Resected Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Docetaxel, Bevacizumab, and Erlotinib Versus Chemotherapy Alone in Resected NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 142; US_IST_12218; AVF3923s
Record Dates: First submitted 2007-12-26; First posted 2008-02-22 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Resected; Carboplatin; Docetaxel; Bevacizumab; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel/Carboplatin/Bevacizumab/Erlotinib (Experimental)
  Interventions: Drug: Docetaxel/Carboplatin/Bevacizumab/Erlotinib
- Docetaxel and Carboplatin (Active Comparator)
  Interventions: Drug: Docetaxel/Carboplatin

INTERVENTIONS:
Drug: Docetaxel/Carboplatin/Bevacizumab/Erlotinib — Docetaxel 75mg/m2 IV D1 Carboplatin AUC=6 IV D1 Bevacizumab 15mg/kg IV D1
  Docetaxel should be administered before carboplatin.
  After completion of four cycles of treatment, patients in Cohort A will then proceed with Maintenance treatment defined as follows:
  Maintenance Treatment for patients in Cohort A:
  Bevacizumab 15mg/kg IV D1 Erlotinib 150mg PO daily
  Treatment cycle = 21 days. Patients will complete 8 cycles (24 weeks) of maintenance therapy unless there is evidence of disease recurrence or unacceptable toxicity.
  Arms: Docetaxel/Carboplatin/Bevacizumab/Erlotinib
Drug: Docetaxel/Carboplatin — Adjuvant Treatment Cohort B:
  Docetaxel 75mg/m2 IV D1 Carboplatin AUC=6 IV D1
  Docetaxel should be administered before carboplatin.
  Treatment cycle = 21 days. Patients in Cohort B will complete 4 cycles of treatment.
  Arms: Docetaxel and Carboplatin

SUMMARY:
Multicenter randomized phase II trial to examine the safety and efficacy of carboplatin, docetaxel, bevacizumab followed by maintenance bevacizumab and erlotinib in patients with completely resected stage IB, II, and select III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-confirmed non-small cell lung cancer (adenocarcinoma, squamous, large cell and undifferentiated). Mixed small cell and non-small histologies are excluded.
2. Patients with completely resected (R0) stage IB, II, and select III NSCLC. The following stages are eligible:

   IB T2 N0 IIA T1 N1 IIB T2 N1 IIB T3 N0 IIIA T3 N1
   * Bronchioalveolar carcinoma that presents as a single, solitary discrete nodule or mass may be included
   * Patients determined to have N2 disease, that was not apparent radiologically preoperatively (and completely resected) can be included.
3. Complete surgical resection defined as the appropriate pulmonary parenchymal resection including lobectomy, bilobectomy, sleeve lobectomy, and pneumonectomy with histologically confirmed negative bronchial margins. Patients treated by segmentectomy or wedge resection are not eligible for this study. Additionally all patients must have had either a mediastinal node dissection or at least, sampling of 2 mediastinal nodal stations (levels 4,7,and 9 for right-sided tumors, and levels 5,6,7, and 9 for left-sided tumors are suggested.)
4. No evidence of metastatic disease
5. ANC >= 1500, platelets >= 100,000 and hemoglobin >= 10.0.
6. Total bilirubin <= ULN. AST and ALT and alkaline phosphatase must be WNL
7. Serum creatinine <= 1.5mg/dl (If greater than 1.5, the creatinine clearance, calculated according to the Cockroft-Gault formula, must be >= 50ml/min).
8. Patients may have had no previous chemotherapy, radiation therapy, angiogenesis inhibitor, or tyrosine kinase inhibitor for non-small cell lung cancer.
9. Patients must be able to understand the nature of this study and give written informed consent.
10. Age >= 18 years
11. Ability to start treatment between 8 and 12 weeks following surgery.
12. Ability to take oral medication.

Exclusion Criteria:

1. Patients with preoperative radiologic evidence of N2 disease by either PET or CT scan (i.e. radiological evidence of metastasis to ipsilateral mediastinal and subcarinal nodes) that is confirmed as N2 disease histologically are excluded. - PLEASE SEE EXCEPTION in section 3.1.2 of protocol
2. Mixed small cell and non-small cell histologies
3. Pulmonary carcinoid tumors
4. Positive bronchial margins
5. History of prior malignancy within 5 years with the exception of skin cancer or cervical carcinoma in situ.
6. Women who are pregnant (positive pregnancy test) or breast-feeding. Subjects of childbearing potential or with partners of childbearing potential (women and men) must use effective birth control measures during treatment.
7. Treatment with a non-approved or investigational drug within 30 days before day 1 of trial treatment.
8. Patients with seizures not controlled with standard medical therapy.
9. Patients with active infection requiring parenteral antibiotics
10. Patients who have had major surgical procedure, open biopsy, or significant traumatic injury within 8 weeks of beginning study treatment or anticipation of need for major surgical procedure during the course of the study
11. Fine needle aspiration, core biopsy or other minor surgical procedure (excluding placement of a vascular access device) within 7 days of beginning study treatment.
12. Patients receiving thrombolytic therapy within 10 days of starting study treatment are also ineligible. Patients may receive prophylactic anticoagulation therapy, 1 mg coumadin daily for port clot prophylaxis.
13. Patients with proteinuria at screening as demonstrated by either:

    * Urine protein creatinine (UPC) ratio >= 1.0 at screening OR
    * Urine dipstick for proteinuria >= 2+ (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate >= 1 g of protein in 24hours to be eligible).
14. Patients with serious nonhealing wound, ulcer, or bone fracture.
15. Patients with evidence of bleeding diathesis or coagulopathy.
16. Patients with history of hemoptysis defined as bright red blood of ½ teaspoon or more per episode) within 8 weeks prior to study treatment.
17. History of myocardial infarction or unstable angina within 6 months of beginning study treatment.
18. Inadequately controlled hypertension (defined as systolic blood pressure > 150 and /or diastolic blood pressure > 100 mmHg on antihypertensive medications).
19. New York Heart Association (NYHA) grade II or greater CHF.
20. Serious cardiac arrhythmia requiring medication.
21. Symptomatic peripheral vascular disease.
22. History of stroke or transient ischemic attack within 6 months prior to beginning bevacizumab.
23. Any prior history of hypertensive crisis or hypertensive encephalopathy.
24. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning study treatment.
25. ECOG Performance status > 1.
26. Peripheral neuropathy> grade 1.
27. Known hypersensitivity to any component of study drugs including platinum or to drugs formulated with polysorbate 80.
28. Impaired oral absorption.
29. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-12; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (26):
- United States (26):
  - Northeast Alabama Medical Center, Anniston, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - RHHP/Hope Cancer Center, Terre Haute, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Jackson Oncology Associates, Jackson, Mississippi
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Adjuvant Treatment
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Started | 55 | 57
Completed | 52 | 47
Not Completed | 3 | 10
Period: Maintenance Treatment
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Started | 49 (3 patients came off study between the end of adjuvant therapy and the start of maintenance) | 0 (Per protocol, only the Docetaxel/Carboplatin/Bevacizumab/Erlotinib arm enters maintenance therapy)
Completed | 34 | 0
Not Completed | 15 | 0

BASELINE CHARACTERISTICS:
Population: All patients on-study
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 79] | 64 [48 to 87] | 64 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants]
  United States | 55 | 57 | 112

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: The length of time, in months, that patients were alive from the end of their treatment without any signs or symptoms of their disease.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Number analyzed (Participants) | 55 | 57
months | NA [NA to NA] — Median DFS cannot be calculated for this arm - not enough participants with events required for this calculation | 55.1 [32.9 to NA] — Upper bound of 95% CI cannot be calculated for this arm

2. Secondary Outcome: Safety
Description: Adverse Events occuring in >15% of patients
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Number analyzed (Participants) | 55 | 57
participants
  Fatigue | 37 | 41
  Nausea | 32 | 36
  Diarrhea | 26 | 24
  Anemia | 18 | 28
  Neutrophil count decreased | 20 | 26
  White blood cell decreased | 18 | 27
  Alopecia | 21 | 21
  Pain | 23 | 15
  Platelet count decreased | 13 | 20
  Constipation | 14 | 18
  Dyspnea | 14 | 17
  Anorexia | 12 | 18
  Hyperglycemia | 18 | 11
  Dysgeusia | 12 | 14
  Mucositis | 12 | 12
  Vomiting | 10 | 13
  Cough | 12 | 8
  Peripheral sensory neuropathy | 15 | 2

3. Secondary Outcome: 2-year Survival
Description: Proportion of patients known to still be alive 2 years after coming on study
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Number analyzed (Participants) | 55 | 57
percentage of participants | 78.2 | 71.9

4. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Number analyzed (Participants) | 55 | 57
months | NA [NA to NA] — Median OS cannot be calculated for this arm - not enough participants with events required for this calculation | NA [NA to NA] — Median OS cannot be calculated for this arm - not enough participants with events required for this calculation

ADVERSE EVENTS:
Arm/Group | Docetaxel/Carboplatin/Bevacizumab/Erlotinib | Docetaxel and Carboplatin
Serious Adverse Events (participants affected / at risk) | 14/55 | 14/57
Other Adverse Events (participants affected / at risk) | 53/55 | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Carboplatin/Bevacizumab/Erlotinib (N=55) | Docetaxel and Carboplatin (N=57)
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bone infection (Infections and infestations) | 0 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Gastrointestinal disorders - Other, hemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatobiliary disorders - Other, cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, haemophilus influenza (Infections and infestations) | 0 | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 | 0
Infections and infestations - Other, pseudomona bacteremia (Infections and infestations) | 1 | 0
Infections and infestations - Other, unspecified (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Carboplatin/Bevacizumab/Erlotinib (N=55) | Docetaxel and Carboplatin (N=57)
Fatigue (General disorders) | 37 | 41
Nausea (Gastrointestinal disorders) | 32 | 36
Diarrhea (Gastrointestinal disorders) | 26 | 24
Anemia (Blood and lymphatic system disorders) | 18 | 28
Neutrophil count decreased (Investigations) | 20 | 26
White blood cell decreased (Investigations) | 18 | 27
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 21
Pain (General disorders) | 23 | 15
Platelet count decreased (Investigations) | 13 | 20
Constipation (Gastrointestinal disorders) | 14 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Anorexia (Metabolism and nutrition disorders) | 12 | 18
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 11
Dysgeusia (Nervous system disorders) | 12 | 14
Mucositis (Gastrointestinal disorders) | 12 | 12
Vomiting (Gastrointestinal disorders) | 10 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 2
Proteinuria (Renal and urinary disorders) | 13 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 7
Fever (General disorders) | 7 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 7 | 5
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 5 | 5
General disorders and administration site conditions - Other, hemorrhage (General disorders) | 7 | 3
Hypertension (Vascular disorders) | 6 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 | 3
Headache (Nervous system disorders) | 4 | 4
Musculoskeletal and connective tissue disorders - Other, body ache (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Infections and infestations - Other, unknown (Infections and infestations) | 1 | 6
Weight loss (Investigations) | 4 | 3
Allergic reaction (Immune system disorders) | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Respiratory, thoracic and mediastinal disorders - Other, unknown (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites